CLINICAL TRIAL: NCT07282431
Title: Clinical Effectiveness of Extracorporeal Shock Wave Therapy Combined With Exercise in Patients With Lateral Epicondylitis
Brief Title: Shockwave Therapy Plus Exercise for Lateral Epicondylitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, salih tan, Doctorate, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MST-1
Record Dates: First submitted 2025-11-16; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Lateral Epicondylitis
Keywords: Lateral epicondylitis Extracorporeal Shock Wave Therapy
MeSH Terms: conditions — Tennis Elbow | interventions — Extracorporeal Shockwave Therapy; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Participants will be randomly assigned to two groups; one group will receive exercise therapy alone,
  Interventions: Other: exercise therapy
- Extracorporeal Shock Wave Therapy (ESWT) (Experimental): Participants will be randomly assigned to two groups; one group will receive exercise therapy alone, while the other group will receive exercise plus Extracorporeal Shock Wave Therapy (ESWT). Clinical efficacy will be assessed by pre- and post-treatment measurements.
  Interventions: Other: Extracorporeal Shock Wave Therapy (ESWT)

INTERVENTIONS:
Other: Extracorporeal Shock Wave Therapy (ESWT) — Extracorporeal Shock Wave Therapy (ESWT)
  Arms: Extracorporeal Shock Wave Therapy (ESWT)
Other: exercise therapy — exercise therapy
  Arms: Control Group

SUMMARY:
The primary objective of this study is to compare the clinical effectiveness of exercise therapy alone versus exercise combined with Extracorporeal Shock Wave Therapy (ESWT) in individuals with lateral epicondylitis, focusing on changes in pain, grip strength, functional status, and overall treatment success.

DETAILED DESCRIPTION:
This randomized, controlled, prospective clinical trial aims to compare the effectiveness of exercise therapy alone versus exercise therapy combined with Extracorporeal Shock Wave Therapy (ESWT) in individuals diagnosed with lateral epicondylitis. The study is conducted at a single center and includes adult participants who meet predefined eligibility criteria.

Participants are randomly assigned to one of two groups: an exercise-only group and an exercise-plus-ESWT group. Both groups follow a 4-week treatment program consisting of 12 sessions delivered three times per week. The exercise program includes isometric, isotonic, and stretching exercises targeting wrist extensors and related musculature. These exercises are demonstrated and supervised by physiotherapists, with participants encouraged to continue them as a home program.

In the intervention group, ESWT is administered once weekly for a total of four sessions. A radial-type ESWT device is used with preset parameters (2.0 bar pressure, 10 Hz frequency, 2000 pulses per session). All ESWT applications are performed by trained physiotherapists.

Clinical assessments occur at baseline and at the end of the 4-week intervention. Pain intensity, upper-extremity functional capacity, and condition-specific functional limitations are measured using validated outcome tools. Global improvement is also recorded at post-treatment to evaluate the participant's perceived benefit.

This study is designed to provide comparative data on the added value of ESWT when combined with a structured exercise program for the management of lateral epicondylitis, with the goal of informing clinical decision-making and optimizing treatment strategies.

ELIGIBILITY:
Inclusion Criteria: Individuals with the following characteristics will be included in the study:

* Being 18 years of age or older
* Having a clinical diagnosis of lateral epicondylitis
* Not having received any other similar treatment within the last 6 months
* Having the cognitive ability to understand the Turkish questionnaire and assessment forms
* Voluntarily agreeing to participate in the study and providing written informed consent

Exclusion Criteria: Individuals with one or more of the following conditions will be excluded from the study:

* Having a history of concomitant systemic, rheumatological, or inflammatory diseases that could affect pain
* Having a history of trauma, surgery, or neurological disease in the upper extremity
* Presence of conditions other than lateral epicondylitis, such as tendinopathy, bursitis, or nerve entrapment
* Having major psychiatric disorders that could affect the pain threshold (e.g., major depression, schizophrenia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Extracorporeal Shock Wave Therapy (ESWT) applied in addition to exercise does not create a significant difference in pain level, grip strength and functional status in individuals with lateral epicondylitis compared to exercise alone. | 8 week
  Pain Intensity (Visual Analog Scale - VAS) Description: Pain intensity will be assessed using the Visual Analog Scale, a 10-cm line ranging from 0 (no pain) to 10 (worst imaginable pain). Participants will mark their perceived pain level on the line.
  Time Frame: Baseline and 8 weeks Outcome Type: Continuous Interpretation: Higher scores indicate worse pain.
Upper Extremity Function (Quick Disabilities of the Arm, Shoulder and Hand Questionnaire - QuickDASH) | 8 week
  Upper Extremity Function (Quick Disabilities of the Arm, Shoulder and Hand Questionnaire - QuickDASH) Description: Functional status will be measured using the QuickDASH questionnaire. Scores range from 0 (no disability) to 100 (severe disability).
  Time Frame: Baseline and 8 weeks Outcome Type: Continuous Interpretation: Higher scores indicate worse functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Salih tan, doctorate, Study Director — Medipol University
Locations (1):
- Istanbul medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No